CLINICAL TRIAL: NCT02255032
Title: A Randomized, Masked, Multicenter Study to Assess the Safety and Efficacy of CLS-TA, Triamcinolone Acetonide Injectable Suspension in the Treatment of Subjects With Macular Edema Following Uveitis
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide in Subjects With Macular Edema Following Non-Infectious Uveitis
Acronym: DOGWOOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS1001-201
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Uveitis; Macular Edema; Uveitis, Posterior; Uveitis, Anterior; Panuveitis; Uveitis, Intermediate
Keywords: uveitis; macular edema; UME; posterior uveitis; anterior uveitis; panuveitis; intermediate uveitis; noninfectious uveitis; triamcinolone acetonide; suprachoroidal space; injection; microneedle; intravitreal injection; corticosteroid; CME; choroid; retina; microinjection; SCS
MeSH Terms: conditions — Uveitis; Macular Edema; Uveitis, Posterior; Uveitis, Anterior; Panuveitis; Uveitis, Intermediate; Choroidal Effusions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 mg CLS-TA (Experimental): Single unilateral, suprachoroidal injection of 40 mg/mL (4 mg in 100 µL) of CLS-TA
  Interventions: Drug: 4 mg CLS-TA
- 0.8 mg CLS-TA (Experimental): Single unilateral, suprachoroidal injection of 8 mg/mL (0.8 mg in 100 µL) of CLS-TA
  Interventions: Drug: 0.8 mg CLS-TA

INTERVENTIONS:
Drug: 4 mg CLS-TA — 40 mg/mL CLS-TA, Clearside's formulation of TA (CLS-TA, triamcinolone acetonide injectable suspension)
  Arms: 4 mg CLS-TA
Drug: 0.8 mg CLS-TA — 8 mg/mL CLS-TA, Clearside's formulation of TA (CLS-TA, triamcinolone acetonide injectable suspension)
  Arms: 0.8 mg CLS-TA

SUMMARY:
The study is designed to evaluate the safety and efficacy of triamcinolone acetonide, CLS-TA, in subjects with macular edema following non-infectious uveitis. A single suprachoroidal injection of one of two doses of CLS-TA will each be evaluated in subjects with macular edema following non-infectious uveitis.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, masked, multicenter study to assess the safety and efficacy of two different doses of CLS-TA in the treatment of subjects with macular edema following non-infectious uveitis. Each subject will receive a single suprachoroidal injection of CLS-TA.

The subjects enrolled in this study will be chosen from subjects with macular edema following non-infectious uveitis. A single injection will be administered via the Clearside microinjector into the suprachoroidal space. The dose injected will either be 4 mg or 0.8 mg of CLS-TA in a total volume of 100 μL. The dose they receive will depend on what their randomization code dictates.

Subjects will be monitored for safety and efficacy for approximately 8 weeks following treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of noninfectious uveitis
* diagnosis of macular edema associated with noninfectious uveitis

Exclusion Criteria:

* any ocular trauma within the immediate 6 months prior to treatment
* any photocoagulation or cryotherapy in the 6 months prior to treatment
* any IVT injection of anti-VEGF treatment in the 2 months prior to treatment
* any eye diseases other than uveitis and ME that could compromise central visual acuity
* any previous suprachoroidal injection of triamcinolone acetonide in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical, Inc.
Locations (11):
- United States (11):
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Waltham, Massachusetts
  - Omaha, Nebraska
  - New York, New York
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 4 mg CLS-TA: Single unilateral, suprachoroidal injection of 40 mg/mL (4 mg in 100 µL) of CLS-TA
  4 mg CLS-TA: 4 mg/mL CLS-TA, Clearside's formulation of TA (CLS-TA, triamcinolone acetonide injectable suspension)
- 0.8 mg CLS-TA: Single unilateral, suprachoroidal injection of 8 mg/mL (0.8 mg in 100 µL) of CLS-TA
  0.8 mg CLS-TA: 0.8 mg/mL CLS-TA, Clearside's formulation of TA (CLS-TA, triamcinolone acetonide injectable suspension)
Period: Overall Study
Arm/Group | 4 mg CLS-TA | 0.8 mg CLS-TA
Started | 17 | 5
Completed | 17 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat set includes all randomly assigned subjects who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg CLS-TA | 0.8 mg CLS-TA | Total
Number analyzed (Participants) | 17 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 17
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (19.65) | 51.8 (16.87) | 52.1 (18.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 9 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 17 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Subfield Thickness, Measured Using Optical Coherence Tomography, After Treatment With CLS-TA in Subjects With Macular Edema Following Uveitis
Time Frame: 2 months
Population: Intent-to-Treat set includes all randomly assigned subjects who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | 4 mg CLS-TA | 0.8 mg CLS-TA
Number analyzed (Participants) | 16 | 5
Microns | -164.44 (173.148) | -78.20 (121.890)
Statistical Analysis 1: Comparison: 4 mg CLS-TA; A paired t-test was used to assess the statistical significance of the change between Baseline and Month 2. A sample size of 16 subjects would have 80% power to detect a difference of 75, assuming a standard deviation of 100, using a paired t-test with a 0.050 two-sided significance level; Test type: Superiority; p = 0.0017, Paired t-test, two-sided — The primary analysis of the primary efficacy endpoint was the comparison between the Baseline and Month 2 values for the 4 mg treatment group. No adjustments for multiplicity were necessary; Mean Difference (Final Values) = -164.44, 95% CI 2-sided [-256.7 to -72.2], Standard Deviation 173.148

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | 4 mg CLS-TA | 0.8 mg CLS-TA
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/5
Other Adverse Events (participants affected / at risk) | 14/17 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg CLS-TA (N=17) | 0.8 mg CLS-TA (N=5)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg CLS-TA (N=17) | 0.8 mg CLS-TA (N=5)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Anterior chamber cell (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Anterior chamber inflammation (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Blindness transient (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 2 (2) — #Study eye
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Conjunctival oedema (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Dry eye (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Dry eye (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Eye pain (Eye disorders) | 3 (3) | 0 (0) — #Study eye
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Keratitis (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Macular oedema (Eye disorders) | 0 (0) | 3 (3) — #Study eye
Macular oedema (Eye disorders) | 2 (2) | 1 (1) — #Fellow eye
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Uveitis (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Uveitis (Eye disorders) | 3 (3) | 0 (0) — #Fellow eye
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Injection site pain (General disorders) | 1 (1) | 1 (1) — #Study eye
Papillitis (General disorders) | 1 (1) | 0 (0) — #Study eye
Papillitis (General disorders) | 1 (1) | 0 (0) — #Fellow eye
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) — #Study eye
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) — #Fellow eye
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of Clearside.